CLINICAL TRIAL: NCT07104539
Title: Strength Training Response of Muscle in GLP-1 Users
Acronym: STRONG-GLP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-707
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Muscle Mass
Keywords: Weight loss; GLP-1 agonist; Obesity; Lean mass; Body composition; Strength training
MeSH Terms: conditions — Weight Loss; Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strenth Training (Experimental): Participants will undergo strength training 3 times per week for 14 weeks.
  Interventions: Behavioral: Strength Training
- Waitlisted control (Other): Participants will have no strength training intervention for 14 weeks. Participants will be offered the same 14-week strength training program after the initial 14 weeks.
  Interventions: Other: Wait first, then strength training

INTERVENTIONS:
Behavioral: Strength Training — Participants taking a GLP-1 will undergo a 14-week strength training regimen to determine changes in muscle mass. They will perform a series of resistance training exercises supervised by a personal trainer on 3 days per week.
  Arms: Strenth Training
Other: Wait first, then strength training — Participants will be waitlisted and receive the 14-week strength training intervention at the end of the waitlist period. During the waitlist period, participants will get no intervention and then be offered the strength training intervention after the first 14 weeks.
  Arms: Waitlisted control

SUMMARY:
GLP-1 medication is being prescribed for weight loss. However, GLP-1 medication may adversely affect muscle mass and muscle function. Moreover, any loss of muscle mass or muscle function with GLP-1 treatment may impair balance and increase fall risk. This is a particular concern among older adults already susceptible to the common muscle strength and muscle function loss with age, yet there is little evidence among this population. This study will address a gap in knowledge regarding the effects of GLP-1 treatment on muscle mass, muscle function, and balance/fall risk among adults age 50 and older.

ELIGIBILITY:
Inclusion Criteria:

* Age, 50y+
* Be taking GLP-1 medicine (Weygovy or Zepbound) for 1 month or less
* Weight <300 lb
* Pass a health and exercise readiness screening

Exclusion Criteria:

* Age <50
* Weight >300 lb
* Osteoporosis
* Active metabolic, neoplastic, or cardiovascular disease
* Unable or unwilling to provide consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Muscle mass by d3-creatine dilution | Water containing creatine isotope consumed in lab; Urine sample collection on Day 0 and Day 3 at baseline and 14 weeks.
  Participants will collect a urine sample prior to be provided a creatine capsule containing 30 milligrams of a naturally-occurring creatine isotope. A glass of water will be provided to wash it down. Participants will be asked to return ~3 days later to provide another urine sample. Urine samples will be analyzed at an off-site laboratory to determine changes in d3-creatine excretion before and after the 14-week strength training intervention.
Balance testing - Percentage of failed recoveries | 2-hour testing session in lab at baseline and 14 weeks.
  Participants will stand on the treadmill with the belt stationary. The belt will then suddenly change to a speed specified by the investigator, and the participant will attempt to step to maintain their balance and establish a stable gait. In addition to the treadmill itself, this system includes an integrated fall arrest harness that is anchored to an overhead gantry that is fixed to the treadmill. This harness prevents any body part but the feet from impacting the treadmill in the event that the participant is unable to maintain their balance after a sudden change in speed.

SECONDARY OUTCOMES:
Muscle function | 500-meter timed walk in lab at baseline and 14 weeks
  Participants will walk 500 meters down and back along a hallway at a self-selected pace. The walk will be measured, supervised, and timed by lab personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Davy, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States